CLINICAL TRIAL: NCT00901472
Title: Sleep Disordered Breathing and Blood Glucose Control in Type 2 Diabetes
Brief Title: Sleep Disordered Breathing and Diabetes
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: #14903B
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes; Obstructive Sleep Apnea
Keywords: Type 2 diabetes,; obstructive sleep apnea
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood was taken for HbA1C
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable type 2 Diabetes (ST2D): Adults with Type 2 diabetes who receive medical care at the University of Chicago

SUMMARY:
The hypothesis of this study is: sleep disordered breathing (SDB), specifically, obstructive sleep apnea, is associated with poorer glucose in the existing type 2 diabetic condition.

In an exploration of this hypothesis, the investigators hope to provide evidence linking SDB to increased severity of disease in the type 2 diabetic patient. By doing so, the investigators ultimately seek to support investigating the use of SDB interventions as an additional method of care in the treatment of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* adult female and male patients with type 2 diabetes who are followed by University of Chicago physicians

Exclusion Criteria:

* patients with the diagnosis of type 1 diabetes (DM); newly diagnosed Type 2 DM patients
* patients with the diagnosis of OSA using CPAP for either 4 or more hours per night or 5 nights per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with type 2 diabetes who are followed by University of Chicago physicians in the endocrinology or primary care clinic will self-identify themselves for participation in response to flyers posted at the check-in desk.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Improvement in glucose tolerance | Day 1 to day 10.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States